CLINICAL TRIAL: NCT00833508
Title: Effect of Preoperative Chemoradiotherapy on Exercise Capacity as Measured by Cardiopulmonary Exercise Testing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 08/H0712/117
Record Dates: First submitted 2009-01-30; First posted 2009-02-02 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2016-02

CONDITIONS: Colorectal Cancer
Keywords: Exercise capacity; Chemoradiotherapy; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Test arm (Experimental): Patients undergoing preoperative chemoradiotherapy will have their exercise capacity measured before and after chemoradiotherapy.
  Interventions: Other: Cardiopulmonary exercise testing

INTERVENTIONS:
Other: Cardiopulmonary exercise testing — Cardiopulmonary exercise testing involves cycling on an exercise bicycle whilst oxygen consumption and carbon dioxide generation are measured from expired gases. This is used to calculate patient fitness from their peak oxygen consumption and their anaerobic threshold.

SUMMARY:
This study will investigate the effect of preoperative chemoradiotherapy on exercise capacity as measured by cardiopulmonary exercise testing in patients with colorectal cancer.

DETAILED DESCRIPTION:
Chemoradiotherapy is associated with adverse effects. Patients with certain colorectal cancers undergo chemoradiotherapy prior to surgical resection. We intend to assess patient exercise capacity before and after chemoradiotherapy to assess whether this deteriorates. If there is a deleterious effect, this may affect operative outcome.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 65
* Colorectal cancer requiring preoperative chemoradiotherapy

Exclusion Criteria:

* Inability to walk, or exercise on a bicycle or treadmill
* Inability to understand instructions for CPET testing
* ASA grade 4 or 5 (indicating severe cardiovascular co-morbidity and not expected to survive surgery)
* Contraindications to Exercise Testing
* Myocardial infarction occurring 10 days or less before CPX testing
* Symptomatic arrythmias
* Left Main Stem coronary disease of >50%
* Severe hypertension (SBP>180mmHg)
* Resting SpO2 <85%
* Acute cardiac inflammatory conditions (myocarditis, pericarditis)
* Unstable angina with symptoms within 4 days
* Dissecting aneurysm of aorta
* Acute pyrexial illness
* Thyrotoxicosis
* Syncopal episodes
* Lower limb thrombosis (arterial or venous)

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-01; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Change of Anaerobic threshold of 1.5ml/min/kg or more | 6 weeks

SECONDARY OUTCOMES:
Operative outcome | 6-10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Stonell, FRCA MBBCh, Principal Investigator — Imperial NHS Trust at St Mary's Hospital
Locations (1):
- Imperial NHS Trust, St Mary's Hospital, Praed Street, London, United Kingdom

REFERENCES:
- [Background] Older P, Smith R, Courtney P, Hone R. Preoperative evaluation of cardiac failure and ischemia in elderly patients by cardiopulmonary exercise testing. Chest. 1993 Sep;104(3):701-4. doi: 10.1378/chest.104.3.701. PMID 8365279